CLINICAL TRIAL: NCT00506922
Title: Phase I/II Study of Pentostatin Combined With Tacrolimus and Mini-Methotrexate for GVHD Prevention After Matched-Unrelated Donor Blood and Marrow Transplantation
Brief Title: Phase I/II Study of Pentostatin Combined With Tacrolimus and Mini-Methotrexate for GVHD Prevention After MUD BMT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID00-132
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Results first posted 2011-03-28 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2012-08

CONDITIONS: Leukemia; Lymphoma
Keywords: Graft-Versus-Host Disease; GVHD Prevention; Hodgkin's Disease; Leukemia; Lymphoma; Methotrexate; Tacrolimus; Pentostatin
MeSH Terms: conditions — Leukemia; Lymphoma; Graft vs Host Disease; Hodgkin Disease | interventions — Pentostatin; Tacrolimus; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- No Pentostatin (Experimental): Group 1: No Pentostatin
  Interventions: Drug: Pentostatin; Drug: Tacrolimus; Drug: Methotrexate
- Pentostatin 0.5 (Experimental): Group 2: Pentostatin 0.5 mg/m^2
  Interventions: Drug: Pentostatin; Drug: Tacrolimus; Drug: Methotrexate
- Pentostatin 1 (Experimental): Group 3: Pentostatin 1 mg/m^2
  Interventions: Drug: Pentostatin; Drug: Tacrolimus; Drug: Methotrexate
- Pentostatin 1.5 (Experimental): Group 4: Pentostatin 1.5 mg/m^2
  Interventions: Drug: Pentostatin; Drug: Tacrolimus; Drug: Methotrexate
- Pentostatin 2 (Experimental): Group 5: Pentostatin 2 mg/m^2
  Interventions: Drug: Pentostatin; Drug: Tacrolimus; Drug: Methotrexate

INTERVENTIONS:
Drug: Pentostatin — Given intravenously on days +8, +15, +22 and +30 post transplant:
  Group 2 - Pentostatin 0.5 mg/m^2
  Group 3 - Pentostatin 1 mg/m^2
  Group 4 - Pentostatin 1.5 mg/m^2
  Group 5 - Pentostatin 2 mg/m^2
  Other Names: Nipent; Deoxycoformycin; DCF
Drug: Tacrolimus — Given intravenously from day -2, and will be switched to oral dosing when tolerated.
  Other Names: Prograf
Drug: Methotrexate — Given intravenously on days +1, +3, and +6 at the dose of 5 mg/m2.

SUMMARY:
Primary Objective:

1. To determine efficacy of escalating doses of pentostatin in combination with tacrolimus and methotrexate for the prevention of acute graft-versus-host disease (GVHD) in the context of unrelated donor and one antigen mismatched related donor transplantation.

Secondary Objectives:

1. To determine safety of escalating doses of pentostatin in combination with tacrolimus and methotrexate.
2. To reduce the incidence of acute GVHD following transplants with unrelated donor to 40%.
3. To document blood levels of tacrolimus when combined with pentostatin.

DETAILED DESCRIPTION:
During the study, patients will have blood, urine, bone marrow, and X-ray exams done. These exams are done to monitor the results of the transplantation. Blood tests will be done daily while patients are hospitalized.

Patients in this study will receive chemotherapy and/or radiation to treat their malignancy and prevent graft rejection. This is given before the infusion of donor cells.

Patients with myeloid leukemias may receive busulfan by vein (IV) for 4 days and cyclophosphamide by vein for 2 days.

Patients with lymphoid malignancies may receive thiotepa by vein in one dose, cyclophosphamide by vein for 2 days, and irradiation for 4 days.

Other chemotherapy treatments may be used before donor cell infusion.

IV injections will be given through a previously inserted catheter that extends into the vena cava (a large chest vein).

Patients will be randomly picked (as in the toss of a coin) to receive one of five different treatments. This is done to learn the benefit of pentostatin treatment and the appropriate dose. Four of the treatments will use different dose schedules of pentostatin. The fifth treatment group will receive no pentostatin at all. All patients receive tacrolimus and methotrexate.

Pentostatin will be given by vein in 4 doses during the first month after transplant. Tacrolimus (FK506) will be given by vein or mouth for 6 months. Methotrexate will be given by vein for 3 doses in the first week after transplant.

Patients will receive blood and platelet transfusions after the transplant. The number of transfusions will depend on how quickly the blood cell counts return to a normal range.

Patients will remain in the hospital for about 4-6 weeks and in the Houston area for 100 days after the transplant.

This is an investigational study. All of the study drugs are commercially available. Pentostatin will not be used for GVHD prevention outside of this study. A total of 150 patients will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving allogeneic hematopoietic transplants from an unrelated donor or one antigen mismatched related donors.
2. Patients with AML, ALL, Hodgkin's disease, MDS (including CMML), CML in late chronic or accelerated phase or in blast crisis, and lymphoma in first or later relapses.
3. Patients must have bilirubin < 1.5 mg/dL, DLCO > 50% predicted, LVEF > 45% and performance status 0 or 1.
4. Candidates must have a creatinine level < 1.5 mg/dL or a calculated creatinine clearance > 60 ml/min.

Exclusion Criteria:

1. HIV seropositivity
2. Uncontrolled infection
3. Pregnancy
4. Candidates should not have received chemotherapy other than hydroxyurea or Gleevec for at least 3 weeks prior to treatment. Maintenance therapy with oral chemotherapy is acceptable. Treatment day is defined as transplant day +8, which is the date of first dose of pentostatin.
5. Diagnosis of myelofibrosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2000-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcos de Lima, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Parmar S, Del Lima M, Zou Y, Patah PA, Liu P, Cano P, Rondon G, Pesoa S, de Padua Silva L, Qazilbash MH, Hosing C, Popat U, Kebriaei P, Shpall EJ, Giralt S, Champlin RE, Stastny P, Fernandez-Vina M. Donor-recipient mismatches in MHC class I chain-related gene A in unrelated donor transplantation lead to increased incidence of acute graft-versus-host disease. Blood. 2009 Oct 1;114(14):2884-7. doi: 10.1182/blood-2009-05-223172. Epub 2009 Aug 4. PMID 19654407
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: September 15, 2000 to July 26, 2007; All recruitment done at UT MD Anderson Cancer Center
Pre-assignment Details: A total of 150 patients were enrolled, and 147 were available for analysis. Two patients assigned to the 1.5 mg/m^2 arm were removed without receiving treatment (due to ineligibility, and poor donor cell collection). A patient assigned to arm 2.0 mg/m^2 withdrew consent before being treated.
Period: Overall Study
Arm/Group | No Pentostatin | Pentostatin 0.5 | Pentostatin 1 | Pentostatin 1.5 | Pentostatin 2
Started | 37 | 10 | 29 | 63 | 11
Completed | 37 | 10 | 29 | 61 | 10
Not Completed | 0 | 0 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Pentostatin | Pentostatin 0.5 | Pentostatin 1 | Pentostatin 1.5 | Pentostatin 2 | Total
Number analyzed (Participants) | 37 | 10 | 29 | 63 | 11 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 10 | 28 | 61 | 11 | 146
  >=65 years | 1 | 0 | 1 | 2 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (19) | 42 (23) | 47 (20) | 50 (22) | 45 (32) | 46.8 (23.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 3 | 11 | 30 | 7 | 66
  Male | 22 | 7 | 18 | 33 | 4 | 84
Region of Enrollment [Number; unit: participants]
  United States | 37 | 10 | 29 | 63 | 11 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Without GVHD at 100 Days
Description: The primary efficacy endpoint of escalating doses Pentostatin with Tacrolimus + Methotrexate is success, defined to be that the patient is alive, engrafted, and without acute graft-versus-host disease (GVHD) at 100 days.
Time Frame: 100 days
Population: All analysis was intention to treat (ITT).
Measure: Number; unit: participants
Groups:
- Pentostatin: 150 patients were enrolled, 2 patients not treated, 38 patients were Group 1 (no Pentostatin), the remaining Groups 2,3,4 and 5, 110 patients were analysed that received the Pentostatin.
Arm/Group | Pentostatin
Number analyzed (Participants) | 147
participants | 100

ADVERSE EVENTS:
Time Frame: 7 Years
Arm/Group | No Pentostatin | Pentostatin 0.5 | Pentostatin 1 | Pentostatin 1.5 | Pentostatin 2
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/10 | 0/29 | 0/61 | 0/10
Other Adverse Events (participants affected / at risk) | 28/37 | 9/10 | 17/29 | 40/61 | 7/10
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Pentostatin (N=37) | Pentostatin 0.5 (N=10) | Pentostatin 1 (N=29) | Pentostatin 1.5 (N=61) | Pentostatin 2 (N=10)
Increased Creatinine (Renal and urinary disorders) | 11 (11) | 6 (6) | 4 (4) | 21 (21) | 4 (4)
TTP/HUS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 7 (7)
CMV (Infections and infestations) | 21 (21) | 3 (3) | 12 (12) | 27 (27) | 5 (5)
bacterial (Infections and infestations) | 24 (24) | 6 (6) | 17 (17) | 38 (38) | 7 (7)
viral (Infections and infestations) | 5 (5) | 2 (2) | 7 (7) | 24 (24) | 1 (1)
parasite (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
fungal (Infections and infestations) | 5 (5) | 2 (2) | 7 (7) | 24 (24) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No